CLINICAL TRIAL: NCT06653686
Title: Study on the Efficacy and Safety of Extracorporeal High-Frequency Hyperthermia in the Treatment of Refractory Gout
Brief Title: Study on the Efficacy and Safety of Thermotherapy in the Treatment of Refractory Gout
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024JD0925
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Refractory Gout
MeSH Terms: conditions — Gout | interventions — Febuxostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Febuxostat (Active Comparator)
  Interventions: Drug: Febuxostat
- Hyperthermia combined with febuxostat (Experimental)
  Interventions: Other: Hyperthermia combined with oral febuxostat.

INTERVENTIONS:
Other: Hyperthermia combined with oral febuxostat. — Extracorporeal high-frequency hyperthermia combined with oral febuxostat
  Arms: Hyperthermia combined with febuxostat
Drug: Febuxostat — The control group subjects were administered oral febuxostat.
  Arms: Febuxostat

SUMMARY:
Gout is a crystal-related arthropathy caused by purine metabolism disorder or decreased uric acid excretion. It can manifest as acute recurrent arthritis, tophus formation, tophaceous chronic arthritis, and urate nephropathy, with severe cases potentially leading to joint disability, renal insufficiency, and damage to other vital organs.Poor long-term control of uric acid levels may result in the progression of refractory gout in some patients, characterized by persistently elevated serum uric acid levels, recurrent acute arthritis, and multiple or progressive tophi, severely affecting quality of life and imposing a significant economic burden on patients.Currently, clinical research on refractory gout is relatively limited, and both domestic and international guidelines continue to recommend uric acid-lowering therapy to slow disease progression.However, due to poor adherence, intolerance to uric acid-lowering drugs, or dose limitations caused by coexisting chronic kidney disease, achieving target serum uric acid levels in these patients is often difficult, and their clinical symptoms are challenging to alleviate effectively.

In recent years, thermotherapy, as a non-pharmacological treatment modality, has garnered increasing attention for its effects in alleviating chronic pain, promoting blood circulation, and reducing inflammatory responses.Its primary mechanisms include: 1) increasing local temperature to influence the solubility of monosodium urate (MSU) crystals, promoting their dissolution, reducing gout attacks, and accelerating the resolution of gout flares;2) elevated local temperature promotes vasodilation and blood circulation, increasing the supply of oxygen and nutrients, facilitating the clearance of uric acid and inflammatory mediators;3) thermotherapy enhances local immune responses by boosting cellular phagocytic activity; 4) it may act as a stimulus transmitted to the central nervous system alongside pain impulses, disrupting pain transmission pathways and resulting in the attenuation or elimination of pain sensations. In recent years, thermotherapy has been widely used in clinical practice as a non-invasive, adjunctive treatment for various conditions, such as tumors, lumbar disc herniation, chronic prostatitis, pelvic inflammatory disease, endometriosis-associated dysmenorrhea, and osteoarthritis, due to its proven efficacy, non-invasive nature, and minimal adverse effects.A study from China demonstrated that thermotherapy has significant therapeutic effects on patients with acute gout attacks, effectively alleviating acute symptoms and reducing inflammatory responses. In this study, the overall clinical efficacy rate of the treatment group (thermotherapy combined with conventional therapy) was significantly higher at 90.0% compared to 72.5% in the control group. Moreover, on day 1 and day 3 post-treatment, the VAS scores of the treatment group (4.11±0.76, 3.23±0.53) were significantly lower than those of the control group (5.23±1.21, 4.23±0.76), and the treatment group had lower ESR and CRP levels than the control group after treatment (P<0.05).Therefore, the primary aim of this study is to investigate the efficacy of thermotherapy in reducing gout attacks. However, there is currently no large-scale, multicenter clinical research evidence evaluating the clinical effectiveness of thermotherapy in patients with refractory gout.

In summary, considering the critical regulatory role of temperature in the formation and deposition of monosodium urate crystals and the fundamental principles of extracorporeal high-frequency thermotherapy, we hypothesize that extracorporeal high-frequency thermotherapy could reasonably reduce MSU crystal burden, lower uric acid levels, alleviate local inflammation, and decrease the frequency of gout attacks through its thermal effects.This study aims to evaluate the efficacy of extracorporeal high-frequency thermotherapy in patients with refractory gout through a randomized controlled trial, exploring its effects on reducing gout attack frequency, improving uric acid metabolism, and alleviating inflammation. Additionally, the study will assess the impact of thermotherapy on patients' quality of life, physical function, and metabolic parameters, with the goal of providing new effective strategies for the treatment of refractory gout in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old;
2. Meeting the diagnostic criteria for refractory gout, defined as fulfilling at least one of the following three conditions: 1) Blood uric acid remains ≥360 μmol/L despite adequate doses and duration of urate-lowering drugs, either alone or in combination (adequate treatment is defined as single-drug therapy at standard doses for more than 6 months, or maximum doses for more than 3 months, with blood uric acid still ≥360 μmol/L; combination therapy for more than 3 months with blood uric acid still ≥360 μmol/L); 2) More than two gout flares per year despite standardized treatment; 3) Presence of multiple or progressive tophi;
3. History of at least three gouty arthritis flares in the past 12 months prior to enrollment;
4. Understanding the purpose and procedures of the study and providing signed informed consent.

Exclusion Criteria:

1. Acute gout flare within 2 weeks prior to screening;
2. Secondary gout due to hematological diseases, chemotherapy, radiotherapy, renal failure, or medications (e.g., diuretics such as furosemide, torsemide, hydrochlorothiazide, aspirin, niacin [vitamin B3], antituberculosis drugs, immunosuppressants such as cyclosporine);
3. Other secondary joint pain (e.g., joint pain caused by rheumatoid arthritis or systemic lupus erythematosus) or joint pain of unknown cause;
4. Patients with cardiac, pulmonary, hepatic, or renal insufficiency; active tuberculosis; mental illness or consciousness disorders;
5. Patients with bone marrow hematopoietic insufficiency; leukemia; a tendency for major bleeding; or a history of malignant tumors;
6. Polyarticular gouty arthritis involving more than four joints;
7. Presence or suspicion of active or recurrent bacterial, fungal, or viral infections, including tuberculosis, HIV, or hepatitis B or C infections;
8. Allergy to the study drugs; patients with heat insensitivity;
9. Patients currently using mercaptopurine or azathioprine; patients taking CYP3A4 inhibitors or P-gp inhibitors;
10. Major surgery within the last 3 months or unhealed surgical wounds;
11. Presence of stents or metal implants;
12. Local skin lesions or infections;
13. Pregnant or breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The number of gout flares during the treatment period | From enrollment to the end of treatment at 20 weeks

SECONDARY OUTCOMES:
The proportion of patients experiencing ≥1 or ≥2 gout flares during the treatment period | From enrollment to the end of treatment at 20 weeks
The time to the first gout flare during the treatment period | From enrollment to the end of treatment at 20 weeks
Changes in serum uric acid levels by the end of the treatment period | From enrollment to the end of treatment at 20 weeks
  Serum uric acid levels will be measured using Uricase-UV method. The change in uric acid levels from baseline to the end of the treatment period will be analyzed.
Proportion of patients achieving target uric acid levels by the end of the treatment period | From enrollment to the end of treatment at 20 weeks
  The proportion of patients achieving a target serum uric acid level of < 360μmol/L will be calculated at the end of the treatment period, using Uricase-UV method to assess uric acid levels.
Percentage reduction in febuxostat dosage by the end of the treatment period | From enrollment to the end of treatment at 20 weeks
  Percentage reduction in febuxostat dosage by the end of the treatment period, investigating changes in febuxostat dosage in the trial and control groups during the study.
Changes in the volume of monosodium urate (MSU) in target joints by the end of the treatment period | From enrollment to the end of treatment at 20 weeks
Changes in C-reactive protein (CRP) levels by the end of the treatment period | From enrollment to the end of treatment at 20 weeks
  CRP will be measured using the immunoturbidimetric method, and changes from baseline to the end of the treatment period will be evaluated.
Changes in erythrocyte sedimentation rate (ESR) by the end of the treatment period | From enrollment to the end of treatment at 20 weeks
  ESR will be measured using an instrument-based method, and changes from baseline to the end of the treatment period will be assessed.
Changes in TH1/TH2-related cytokines by the end of the treatment period | From enrollment to the end of treatment at 20 weeks
  These cytokines will be measured using flow cytometry, and changes from baseline to the end of the treatment period will be evaluated.
Changes in fasting blood glucose at the end of the treatment period | From enrollment to the end of treatment at 20 weeks
  Fasting blood glucose will be measured using the glucose oxidase method, and the change from baseline to the end of the treatment period will be evaluated.
Changes in lipid levels at the end of the treatment period | From enrollment to the end of treatment at 20 weeks
  Lipid levels (including triglycerides, cholesterol, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol) will be measured using enzymatic methods or homogeneous enzymatic colorimetric methods. The overall change in lipid levels from baseline to the end of the treatment period will be assessed.
Changes in quality of life by the end of the treatment period | From enrollment to the end of treatment at 20 weeks
  Changes in quality of life assessed by the The Short-From-36 Health Survey(SF-36). The SF-36 Physical Functioning Scale ranges from 0 to 100, with higher scores indicating better physical function.
Changes in physical function by the end of the treatment period | From enrollment to the end of treatment at 20 weeks
  Changes in physical function at the end of the treatment period were assessed using the Health Assessment Questionnaire (HAQ) Disability Index.The scale ranges from 0 to 3, with higher scores indicating worse physical function.
Comparison of patient treatment satisfaction at the end of the treatment period. | From enrollment to the end of treatment at 20 weeks
  Patient satisfaction at the end of the treatment period was assessed using the Treatment Satisfaction Questionnaire.The scale ranges from 0 to 28, with higher scores indicating greater satisfaction with the treatment.
Incidence of adverse events | From enrollment to the end of study at 24 weeks